CLINICAL TRIAL: NCT03107819
Title: Plasma and Urine Metabolomics for Biomarker Discovery in Children With Eosinophilic Esophagitis
Brief Title: Metabolomics for Biomarker Discovery in Children With EoE
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Lindsay Marie Moye, MD, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-16-1078
Record Dates: First submitted 2017-03-24; First posted 2017-04-11 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Eosinophilic Esophagitis
Keywords: Plasma metabolomics; Urinary metabolomics; Metabonomics; Biomarker discovery
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral venous blood, urine, esophageal mucosa biopsies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients undergoing EGD: Subjects ages 2-18 years undergoing upper endoscopy (EGD) will submit a blood and urine specimen for plasma and urine metabolomics profiling.
  Interventions: Diagnostic Test: Plasma and urine metabolomics

INTERVENTIONS:
Diagnostic Test: Plasma and urine metabolomics — Through the use of high-pressure liquid chromatography and mass spectrometry, quantitative measurements of targeted metabolites associated with amino acids, methylation, acetylation and the tricarboxylic acid (TCA) cycle will be analyzed on the blood and urine specimens.

SUMMARY:
The investigators are seeking to enroll 8 children ages 2-18 already undergoing upper endoscopy. For the purposes of research, a peripheral blood and clean catch urine specimen will be obtained to measure plasma and urine metabolomics. The data will be used to determine if there are any key differences in the metabolite profile of subjects found to have eosinophilic esophagitis (EoE) versus non-EoE subjects. Once these metabolites are identified, the investigators will seek to enroll many more subjects for a validation phase.

DETAILED DESCRIPTION:
Eosinophilic esophagitis (EoE) is a disorder of the esophagus triggered by food and/or environmental allergens and is characterized by symptoms of esophageal dysfunction and eosinophilia of the esophagus. The standard of care for diagnosing and monitoring EoE is with biopsies of the esophagus. There are currently no known biomarkers that correlate with the inflammatory activity of esophageal mucosa, and patients' symptoms alone are insufficient in providing a reliable assessment. Some studies report that patients with EoE may undergo endoscopy up to 11 times in one year. Finding a non-invasive biomarker would therefore be of high clinical and economic interest.

The investigators will seek to enroll 8 children ages 2-18 years already undergoing esophagogastroduodenoscopy (EGD). For the purposes of research, a peripheral blood specimen will be collected at the same time of peripheral intravenous (IV) placement, which is routinely performed for the purposes of sedation during endoscopy, thereby avoiding extra needle sticks. A urine sample will also be collected on the day of the EGD. These specimens will then be analyzed for plasma and urine metabolomics to evaluate for any derangements in EoE versus non-EoE subjects.

Risks to participants undergoing EGD are the same as they would be if they were not enrolled in the study as no additional biopsies will be taken. Risks associated with a blood draw are minimal and include some discomfort, such as lightheadedness, fainting, bruising, soreness, clotting and bleeding at the site of the needle stick, and in rare cases, infection. Collection of the urine specimen is by clean catch in only toilet-trained individuals.

This study should yield valuable information regarding plasma and urine metabolomics in EoE versus non-EoE subjects. Once this "discovery" data set is analyzed, future research could then focus specifically on those abnormal metabolites and seek to enroll many more subjects for a validation phase.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients, ages 2-18 years, undergoing EGD with biopsies of the esophagus.
2. Children with known EoE will only be enrolled if his/her biopsy on the day of specimen collection demonstrates ≥15 eosinophils (eos) per high power field (hpf).

Exclusion Criteria:

1. Presence of other disorders associated with similar clinical, histological or endoscopic features, such as proton pump inhibitor (PPI)-responsive esophageal eosinophilia, esophageal eosinophilia associated with gastroesophageal reflux, Crohn's disease, infectious esophagitis (i.e. herpes simplex virus or candida), drug-associated esophagitis, collagen vascular disease, hypereosinophilic syndrome and eosinophilic gastroenteritis.
2. Children with known EoE and biopsy demonstrating <15 eos/hpf at the time of specimen collection.
3. Inability to provide a clean catch urine specimen (i.e. not toilet-trained).

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children ages 2-18 years already undergoing upper endoscopy (EGD)
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Plasma and urine metabolomics | baseline
  parts per million

CONTACTS AND LOCATIONS:
Overall Officials: Jon M Rhoads, MD, Study Director — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furuta GT, Liacouras CA, Collins MH, Gupta SK, Justinich C, Putnam PE, Bonis P, Hassall E, Straumann A, Rothenberg ME; First International Gastrointestinal Eosinophil Research Symposium (FIGERS) Subcommittees. Eosinophilic esophagitis in children and adults: a systematic review and consensus recommendations for diagnosis and treatment. Gastroenterology. 2007 Oct;133(4):1342-63. doi: 10.1053/j.gastro.2007.08.017. Epub 2007 Aug 8. PMID 17919504
- [Background] Gupta SK. Noninvasive markers of eosinophilic esophagitis. Gastrointest Endosc Clin N Am. 2008 Jan;18(1):157-67; xi. doi: 10.1016/j.giec.2007.09.004. PMID 18061109
- [Background] Dellon ES, Gonsalves N, Hirano I, Furuta GT, Liacouras CA, Katzka DA; American College of Gastroenterology. ACG clinical guideline: Evidenced based approach to the diagnosis and management of esophageal eosinophilia and eosinophilic esophagitis (EoE). Am J Gastroenterol. 2013 May;108(5):679-92; quiz 693. doi: 10.1038/ajg.2013.71. Epub 2013 Apr 9. PMID 23567357
- [Background] Cianferoni A, Spergel JM. Immunotherapeutic approaches for the treatment of eosinophilic esophagitis. Immunotherapy. 2014;6(3):321-31. doi: 10.2217/imt.14.3. PMID 24762076
- [Background] Schlag C, Miehlke S, Heiseke A, Brockow K, Krug A, von Arnim U, Straumann A, Vieth M, Bussmann C, Mueller R, Greinwald R, Bajbouj M. Peripheral blood eosinophils and other non-invasive biomarkers can monitor treatment response in eosinophilic oesophagitis. Aliment Pharmacol Ther. 2015 Nov;42(9):1122-30. doi: 10.1111/apt.13386. Epub 2015 Aug 27. PMID 26314389
- [Background] Kagalwalla AF, Shah A, Li BU, Sentongo TA, Ritz S, Manuel-Rubio M, Jacques K, Wang D, Melin-Aldana H, Nelson SP. Identification of specific foods responsible for inflammation in children with eosinophilic esophagitis successfully treated with empiric elimination diet. J Pediatr Gastroenterol Nutr. 2011 Aug;53(2):145-9. doi: 10.1097/MPG.0b013e31821cf503. PMID 21788754
- [Background] Molina-Infante J, Arias A, Barrio J, Rodriguez-Sanchez J, Sanchez-Cazalilla M, Lucendo AJ. Four-food group elimination diet for adult eosinophilic esophagitis: A prospective multicenter study. J Allergy Clin Immunol. 2014 Nov;134(5):1093-9.e1. doi: 10.1016/j.jaci.2014.07.023. Epub 2014 Aug 28. PMID 25174868
- [Background] Patti GJ, Yanes O, Siuzdak G. Innovation: Metabolomics: the apogee of the omics trilogy. Nat Rev Mol Cell Biol. 2012 Mar 22;13(4):263-9. doi: 10.1038/nrm3314. PMID 22436749
- [Background] Collino S, Martin FP, Rezzi S. Clinical metabolomics paves the way towards future healthcare strategies. Br J Clin Pharmacol. 2013 Mar;75(3):619-29. doi: 10.1111/j.1365-2125.2012.04216.x. PMID 22348240
- [Background] Zhang A, Sun H, Wang P, Han Y, Wang X. Modern analytical techniques in metabolomics analysis. Analyst. 2012 Jan 21;137(2):293-300. doi: 10.1039/c1an15605e. Epub 2011 Nov 21. PMID 22102985
- [Background] Sarosiek I, Schicho R, Blandon P, Bashashati M. Urinary metabolites as noninvasive biomarkers of gastrointestinal diseases: A clinical review. World J Gastrointest Oncol. 2016 May 15;8(5):459-65. doi: 10.4251/wjgo.v8.i5.459. PMID 27190585
- [Background] Stephens NS, Siffledeen J, Su X, Murdoch TB, Fedorak RN, Slupsky CM. Urinary NMR metabolomic profiles discriminate inflammatory bowel disease from healthy. J Crohns Colitis. 2013 Mar;7(2):e42-8. doi: 10.1016/j.crohns.2012.04.019. Epub 2012 May 22. PMID 22626506
- [Background] Davis VW, Schiller DE, Eurich D, Sawyer MB. Urinary metabolomic signature of esophageal cancer and Barrett's esophagus. World J Surg Oncol. 2012 Dec 15;10:271. doi: 10.1186/1477-7819-10-271. PMID 23241138
- [Background] Jung J, Jung Y, Bang EJ, Cho SI, Jang YJ, Kwak JM, Ryu DH, Park S, Hwang GS. Noninvasive diagnosis and evaluation of curative surgery for gastric cancer by using NMR-based metabolomic profiling. Ann Surg Oncol. 2014 Dec;21 Suppl 4:S736-42. doi: 10.1245/s10434-014-3886-0. Epub 2014 Aug 5. PMID 25092158
- [Background] Qiu Y, Cai G, Su M, Chen T, Liu Y, Xu Y, Ni Y, Zhao A, Cai S, Xu LX, Jia W. Urinary metabonomic study on colorectal cancer. J Proteome Res. 2010 Mar 5;9(3):1627-34. doi: 10.1021/pr901081y. PMID 20121166
- [Background] Bertini I, Calabro A, De Carli V, Luchinat C, Nepi S, Porfirio B, Renzi D, Saccenti E, Tenori L. The metabonomic signature of celiac disease. J Proteome Res. 2009 Jan;8(1):170-7. doi: 10.1021/pr800548z. PMID 19072164